CLINICAL TRIAL: NCT00915642
Title: Overnight Weight Loss, Sleep Structure and the Endocrine System
Brief Title: Overnight Weight Loss and Sleep Structure
Acronym: weightsleep
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Associacao Fundo de Incentivo a Psicofarmcologia (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Walter Andre dos Santos Moraes, AFIP
Other Study IDs: CEP1516/07
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Obesity; Healthy
Keywords: Obesity; Weight loss rate; Sleep; Vigil; Metabolism; Actigraphy; Normal
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Normal volunteers: Volunteers, body mass index 17 to 25
- Obese volunteers: Volunteers body mass index higher than 30

SUMMARY:
The objectives of the present study are:

1. to evaluate if overnight weight loss is dependent on sleep structure assessed by polysomnography;
2. to compare weight loss rate during sleep and awake rest;
3. to compare night weight loss profile of normal and obese volunteers.

DETAILED DESCRIPTION:
Weight loss can be caused by loss of body mass due to metabolism and by water loss as insensible water loss, sweating, or excretion in feces and urine. Eighty-three percent of the total weight loss is due to insensible water loss from airways and skin. Water loss rate varies according to changes in activity and ambient temperature and humidity. Although weight loss during sleep is a well-known phenomenon, there are no studies relating it to sleep structure or any other functions during the distinct sleep stages, particularly SWS and REM sleep. There is evidence suggesting a homeostatic mechanism for weight control in animal models and humans. This mechanism is thought to be dependent on energy intake, energy expenditure, and environmental conditions. The literature suggests that sleep is important for weight homeostasis on a long term since sleep shortage is associated with overweight status, but overnight weight variation had not yet been studied. Considering these facts, we hypothesized that the overnight weight loss rate is not uniform throughout the sleep period. We also intend to compare weight loss rate during sleep and awake rest.

Intervention: Normal and obese volunteers will undergo whole night polysomnography with continuous body weight and temperature register after an adaptation night. After that, volunteers will remain awake resting in bed during the following day for continuous weight and temperature register.

ELIGIBILITY:
Inclusion Criteria:

* normal and obese volunteers

Exclusion Criteria:

* serious medical or neurological condition

Ages: 21 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal and obese volunteers
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-01 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Adaptation polysomnography (first night) followed by experimental polysomnography with continuous body weight register (second night) | 8 hours (first night), 8 hours (second night)

SECONDARY OUTCOMES:
Pletysmography | 1 hour (before second night), 1 hour (after second night), 1 hour (after daytime)
Actigraphy (nighttime, daytime) | 24 hours (second night, daytime following second night)
Skin temperature plot | 8 hours (second night), 8 hours (daytime following second night)
Daytime continuous weight register | 8 hours (daytime period following second night)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Moraes, MD PhD, Principal Investigator — AFIP / UNIFESP; Marco Tulio Mello, PhD, Study Director — AFIP / UNIFESP; Sergio Tufik, MD, PhD, Study Chair — AFIP/ UNIFESP
Locations (1):
- Instituto do Sono / Associacao Fundo de Incentivo a Psicofarmacologia, São Paulo, São Paulo, Brazil